CLINICAL TRIAL: NCT04431115
Title: Levels, Patterns and Correlates of Physical Activity, Sedentary Behaviour and Physical Fitness Profile of Primary School Children in Lagos, Nigeria; Development of a Physical Activity Guideline.
Brief Title: Physical Activity, Sedentary Behaviour and Physical Fitness Profile of Primary School Children in Lagos, Nigeria.
Status: Completed | Type: Observational
Sponsor: University of KwaZulu (Other)
Responsible Party: Principal Investigator, Olusegun O. Ojedoyin, PhD candidate, School of health sciences, University of Kwazulu-Natal, University of KwaZulu
Other Study IDs: OjedoyinO
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Stakeholders: Academic experts, Politicians and officials of state ministries of health and education and teachers.
  1. Interviews will be conducted for academic experts, politicians and officials of state ministries of health and education.
  2. Headteachers and physical education teachers will be administered questionnaires.
  Interventions: Other: Interviews
- Parents: Parents of the primary school children to be recruited for the study. Focus group discussion in a group of 3 of ten in each group.
  Interventions: Other: Interviews
- Primary school children aged 6-12 yrs.: A cross sectional survey of the biographical data, socio economic status, physical activity level through appropriate questionnaires will be done.
  A pedometer will be attached to the waist of each of the participants for a consecutive 7 days to objectively determine the level of their physical activity.
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Interviews — Interviews for stakeholders

SUMMARY:
This research study intends to use a mixed method approach(both qualitative and quantitative) to describe and analyse the levels, patterns, and correlates of physical activity((PA), sedentary behaviour(SB), and physical fitness(PF) profiles of primary school children in Lagos state, Nigeria. The study is in four phases.

DETAILED DESCRIPTION:
Phase1 is a scoping review of literature of the level of compliance of all the countries in sub-saharan Africa to the Global observatory on physical activity(GOPA) recommendation on the minimum level of daily physical activity to reduce incidence of non communicable chronic diseases e.g. hypertension, diabetes, obesity etc.

Phase2 is a concurrent mixed method which will explore parents and other stakeholders awareness, understanding and perspectives on PA,SB, and PF among primary school children in Lagos, Nigeria.

Phase 3 is a cross sectional study which will investigate levels, patterns and correlates among physical activity, sedentary behaviour and physical fitness profile of primary school children in Lagos, Nigeria.

Phase 4 is development of physical activity guideline for primary school children in Lagos, Nigeria.

ELIGIBILITY:
Inclusion Criteria: 1.Must be Primary school children between ages 6 and 12 years in Lagos, Nigeria.

-

Exclusion Criteria:

1. Obvious lower limb musculoskeletal diseases.
2. Normal gait impairment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population are primary school children(6-12 yrs) in public and private schools in Lagos state, Nigeria..
Sampling Method: Non-Probability Sample
Enrollment: 1038 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Youth activity profile(YAP) | About 5 days
  It is a self reported questionnaire. It is a physical activity assessment tool designed to assess children and adolescents' physical activity. it is for children between 10-12 years. Three indices are being measured from YAP. These are physical activity at school index(PASI), Physical activity at home index(PAHI) and Sedentary behaviour index(SBI).It consists of 15 total items each scored on a 5- point scale. A higher overall activity score is reflective of a higher level of physical activity(or a greater amount of sedentary behaviour in the case of the SBI. It is on a 5 point scale with 1 being the minimum and 5 maximum to assess physical activity at school.
Children physical activity questionnaire(CPAQ) | for activities over the past seven days.
  It assess mode, frequency and duration of physical activity and sedentary activities. The no of activities run from 1 to 5. 1 being the minimum while 5 is maximum no of days. throughout all domains over the past 7 days. The more the activities participated in each domain the higher the level of physical activity and the lower the sedentary behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Olusegun O Ojedoyin, Principal Investigator — UKZN; Pragashnie Govender, Study Chair — UKZN; Thayananthee Nadasan, Study Director — UKZN; Michael O Olagbegi, Study Director — UKZN
Locations (1):
- Lagos state primary schools, Lagos, Nigeria